CLINICAL TRIAL: NCT02365363
Title: Pulse EnRiched Food and Exercise Clinical Trials (PERFECT Project): Part 2 - Acute Effects of Pulse Ingredients in Food Products on Aerobic Endurance and Substrate Oxidation During Exercise, as Well as, the Blood Glucose, Insulin, Lactate and Food Intake Response Following an Endurance Exercise Session in Adults - Study 3
Brief Title: PERFECT Project - Part 2 - Study 3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Collaborators: Saskatchewan Pulse Growers (Other); Alberta Pulse Growers (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: B2014:114-6
Record Dates: First submitted 2014-12-17; First posted 2015-02-18 (Estimated); Last update posted 2023-01-23 (Actual); Status verified 2021-04

CONDITIONS: Diabetes Prevention; Obesity Prevention
MeSH Terms: interventions — Pea Proteins

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (6):
- Bagel control (Experimental): 100% wheat flour
  Interventions: Other: Control
- Bagel with pea flour (Experimental): Pea flour (30%)
  Interventions: Other: Pea flour
- Bagel with pea fibre (Experimental): Pea fibre (11g)
  Interventions: Other: Pea fibre
- Bagel w/ pea flour + pea fibre (Experimental): Pea flour (30%) + pea fibre (11g)
  Interventions: Other: Pea flour and pea fibre
- Bagel w/ pea flour + pea protein (Experimental): Pea flour (30%) + pea protein (24g)
  Interventions: Other: Pea flour and pea protein
- Bagel w/ pea flour + pea fibre + pea protein (Experimental): Pea flour (30%) + pea fibre (11g) + pea protein (24g)
  Interventions: Other: Pea flour + pea fibre + pea protein

INTERVENTIONS:
Other: Control — Non pulse ingredient bagel
  Arms: Bagel control
Other: Pea flour — Pulse ingredient bagel
  Arms: Bagel with pea flour
Other: Pea fibre — Pulse ingredient bagel
  Arms: Bagel with pea fibre
Other: Pea flour and pea fibre — Pulse ingredient bagel
  Arms: Bagel w/ pea flour + pea fibre
Other: Pea flour and pea protein — Pulse ingredient bagel
  Arms: Bagel w/ pea flour + pea protein
Other: Pea flour + pea fibre + pea protein — Pulse ingredient bagel
  Arms: Bagel w/ pea flour + pea fibre + pea protein

SUMMARY:
The objectives are to test the acute effects of different bagels containing pulse ingredients on: 1) aerobic endurance and substrate oxidation during exercise 2) response of blood glucose, insulin and appetite to an aerobic exercise session, and 3) food intake two hours following the exercise session. We hypothesize that consumption of bagels containing pulse ingredients 60 minutes before exercise will increase aerobic endurance (lower oxygen consumption), decrease carbohydrate oxidation (greater respiratory quotient), and a reduction in lactate production during compared to the same exercise session following the ingestion of a non-pulse food. We also hypothesize that consumption of bagels containing pulse ingredients will lead to lower blood glucose, insulin, appetite and food intake, suggesting lower calorie compensation, following a 60-minute aerobic exercise session compared to the same exercise session following the ingestion of a non-pulse food.

ELIGIBILITY:
* Normoglycemic (<5.6 mmol/L) and normotensive (systolic blood pressure <140 mm Hg and diastolic blood pressure below < 90 mm Hg)
* BMI of 18.5-29.9 kg/m2

Exclusion Criteria:

* Restrained eaters
* Regularly skip breakfast
* Smokers
* Those who are active (organized activities or athletic training at a high intensity; ≥ 150 min per week of moderate to vigorous physical activity)
* Those on medications that may influence study outcomes or have experienced any gastrointestinal related health conditions/surgeries over the past year
* Those unable to walk for an hour continuously

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2016-10; Primary Completion 2017-12-19 (Actual); Study Completion 2017-12-19 (Actual)

PRIMARY OUTCOMES:
Plasma Glucose and Insulin Concentrations | 0-240
  Measured in blood using intravenous catheter. Glucose will be determined by automated methods using Abbot Spectrum CCX Analyzer, and Insulin will be measured by commercially available RIA kits
Food Intake | 120 min
  Ad-libitum meal
Subjective Appetite | 0-240 min
  Motivation-to-eat VAS questionnaire
Exercise intensity | 60-120 min
  Oxygen consumption measured during exercise at 3 time points

SECONDARY OUTCOMES:
Palatability | 5 and 260 min
  Measured by VAS questionnaire
Physical comfort | 0-240 min
  Measured by VAS questionnaire
Energy/fatigue | 0 - 240 min
  Measured by VAS questionnaire
Heart rate | 60-120 min
  To monitor exercise intensity and give a measure of fatigue (cardiovascular drift)
Lactate concentration | 60-120 min
  Measured before, during, and exercise exercise at 3 time points
Substrate Oxidation | 60-120 min
  Respiratory quotient measured during exercise at 3 time points

CONTACTS AND LOCATIONS:
Overall Officials: Peter JH Jones, PhD, Principal Investigator — University of Manitoba, Richardson Centre for Functional Foods and Nutraceuticals
Locations (1):
- Richardson Centre for Functional Foods and Nutraceuticals, University of Manitoba, Winnipeg, Manitoba, Canada